### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | A Randomized, Double-Blind, Placebo-Controlled,<br>Multicentre Study to Evaluate the Efficacy and Safety of<br>Once-Daily, Intranasal Administration of Fluticasone Furoate<br>Nasal Spray 55µg and 110 µg for 4 Weeks in Chinese<br>Paediatric Subjects Ages 2 to 12 Years with Allergic Rhinitis |
|---|---|---|
| <b>Compound Number</b> | ÷ | GW685698 |
| <b>Effective Date</b> | : | 22-JAN-2018 |

**Description:** The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 201492.

- This RAP is intended to describe the demographic and disease characteristics at baseline, efficacy and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **Author's Name and Functional Area:**

| PPD | | |
|---|---|---|
| Statistician, MacroStat (China) Clinical Research Co., Ltd. | 22-JAN-2018 | E-mail approved |

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | 22-JAN-2018 | E-mail approved |
| Statistician, GSK R&D China | 22 3711 2010 | L man approved |
| PPD | 16-JAN-2018 | E-mail approved |
| Clinical Research Physician, GSK R&D China | 10-JAIN-2016 | E-man approved |
| PPD | 17-JAN-2018 | E-mail approved |
| Senior Programmer, GSK R&D China | 1/-JAIN-2016 | E-man approved |
| PPD | 16-JAN-2018 | E-mail approved |
| Senior Clinical Data Scientist, GSK R&D China | 10-JAIN-2016 | E-man approved |
| PPD | 16-JAN-2018 | E-mail approved |
| Associate Study Manager, GSK R&D China | 10-JAIN-2016 | E-man approved |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | <b>Approval Method</b> |
|---|---|---|
| Associate Director, Statistics & Programming, R&D China | 17-JAN-2018 | E-mail approved |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | RTING & ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 7 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | 8 |
| ^ | | NED ANALYOFO | • |
| 3. | | NED ANALYSES | |
| | 3.1.<br>3.2. | Interim Analyses | |
| | 3.2. | Final Analyses | 9 |
| 4. | ANAL' | YSIS POPULATIONS | 9 |
| | 4.1. | Protocol Deviations | 10 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | 'ENTIONS | 12 |
| 6. | STUD | Y POPULATION ANALYSES | 13 |
| ٥. | 6.1. | | |
| | | • | |
| 7. | | ARY STATISTICAL ANALYSES | |
| | 7.1. | Efficacy Analyses | |
| | | 7.1.1. Overview of Planned Efficacy Analyses | |
| | | 7.1.2. Planned Efficacy Statistical Analyses | 15 |
| 8. | SECO | NDARY STATISTICAL ANALYSES | 16 |
| | 8.1. | Efficacy Analyses | 16 |
| | | 8.1.1. Overview of Planned Efficacy Analyses | |
| | | 8.1.2. Planned Efficacy Statistical Analyses | |
| | 8.2. | Safety Analyses | |
| | | 8.2.1. Overview of Planned Analyses | |
| 9. | OTHE | R STATISTICAL ANALYSES | 20 |
| 10. | REFE | RENCES | 21 |
| 11. | APPE | NDICES | 22 |
| | 11.1. | 11. 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| | | Protocol Population | |
| | | 11.1.1. Exclusions from Per Protocol Population | |
| | | 11.1.2. Exclusions of Data from Per Protocol Analyses | |
| | | 11.1.2.1 Inclusion/exclusion/randomisation Criteria Deviations | |
| | 44- | 11.1.2.2 Programmed or and Manual Checks to Identify Deviations | |
| | 11.2. | Appendix 2: Time & Events | 25 |
| | 44.0 | 11.2.1. Protocol Defined Time & Events <sup>1</sup> | |
| | 11.3. | Appendix 3: Assessment Windows | 27 |
| | 11.4. | Appendix 4: Treatment States and Phases | 2ŏ |


| | 11.4.2. | Treatment | States | 28 |
|---|---|---|---|---|
| | | 11.4.2.1. | Treatment States for Concomitant Medications | |
| | | | Data | |
| | | 11.4.2.2. | Treatment States for AE Data | 28 |
| 11.5. | Appendix | 5: Data Di | splay Standards & Handling Conventions | 30 |
| | 11.5.1. | Study Trea | atment & Sub-group Display Descriptors | 30 |
| | 11.5.2. | Baseline D | efinition & Derivations | 30 |
| | | 11.5.2.1. | Baseline Definitions | 30 |
| | | 11.5.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | 30 |
| | 11.5.3. | | Process & Standards | |
| 11.6. | Appendix | 6: Derived | and Transformed Data | 33 |
| | 11.6.1. | General | | 33 |
| | 11.6.2. | Study Pop | ulation | 33 |
| | 11.6.3. | Safety | | 34 |
| | 11.6.4. | | | |
| 11.7. | Appendix | 7: Premati | ure Withdrawals & Handling of Missing Data | 37 |
| | 11.7.1. | Premature | Withdrawals | 37 |
| | 11.7.2. | | f Missing Data | |
| | | | Handing of Missing Dates | |
| | | | Handling of Partial Dates | 38 |
| | | 11.7.2.3. | Handling of Missing Data for Statistical | |
| | | | Analysis | |
| | | | of Potential Clinical Importance | |
| 11.9. | | | ntre Studies | |
| | | | nation of Covariates, Subgroups & Other Strata | |
| | | | e Comparisons & Multiplicity | 42 |
| 11.12. | | | Checking and Diagnostics for Statistical | |
| | | | Analysis Assumptions | |
| 11.13. | | | viations & Trade Marks | |
| | | | ons | |
| | | | S | |
| 11.14. | | | Data Displays | |
| | | | ay Numbering | |
| | | | mple Shell Referencing | |
| | | | e [Priority] | |
| | | | ulation Tables | |
| | | | ulation Figures | |
| | | | ables | |
| | | • | gures | |
| | | | les | |
| | | | ures | |
| | | | JS | |
| 44 45 | | | istings | |
| 11.15. | Appendix | ( ib. ⊨xamr | ole Mock Shells for Data Displays | 65 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP describes the planned analyses and output to be included in the Clinical Study Report for Protocol 201492. |
| Protocol | This RAP is based on the protocol amendment 2 [(Dated: 15/Jan/2016) of study 201492 (GSK Document No.: 2014N205225_02] and eCRF Version 1.0. |
| Primary<br>Objective | <ul> <li>Establish the efficacy of FFNS 55 μg and 110 μg QD versus vehicle placebo<br/>nasal spray in paediatric subjects (ages 2 to 12 years old) with AR.</li> </ul> |
| Primary<br>Endpoint | <ul> <li>Mean change from baseline over the first 2 weeks treatment period in daily,<br/>reflective total nasal symptom scores (rTNSS) in subjects ages 2 to 12 years<br/>old.</li> </ul> |
| Study<br>Design | This study will be a randomized, double-blind, placebo-controlled, multicentre parallel study. The study will be comprised of screen, run-in period (4 to 14 days), treatment period (28 days) and follow up period (3 to 7 days). |
| | During the study period, all investigators, subjects and GlaxoSmithKline (GSK) personnel remain blinded. |
| | Subjects will be assigned to randomized treatments in a 1:1:1 ratio, in accordance with a computer generated randomization schedule provided by GSK. |
| | • The randomization will be centralized and stratified by age (≥2 to ≤6 years old and >6 to ≤12 years old) and by classification of AR (intermittent vs. persistent) to ensure treatment balance in age groups and AR classification groups for both safety and efficacy assessments. |
| Planned<br>Analyses | All decisions regarding final analysis, as defined in this RAP document, will be made prior to Database Freeze (unblinding) of the study data. |
| Analysis<br>Populations | The All Subjects Enrolled Population comprise of all subjects, for whom a record exists on the study database, including screen/run-in failures and any subject who was not screened but experienced an SAE between the date of informed consent and the planned date of the Screening Visit. This population will be used for reporting subject disposition, reasons for screen/run-in failures, and inclusion, exclusion and randomization criteria deviations and SAEs for non-randomized subjects. |
| | The intent-to-treat (ITT) population is defined as all randomized subjects who received at least one dose of study drug. This population will be the primary analysis population for safety and efficacy analysis. Subjects will be assessed according to the treatment they are randomized to. |
| | <ul> <li>The Subset ITT population (2 to 6 years old) is defined as a subset of ITT population comprising subjects aged ≥2 to ≤6 years old.</li> </ul> |
| | The per-protocol (PP) population is defined as all randomized subjects in ITT population who do not have any full protocol deviations. This population will be |

| Overview | Key Elements of the RAP |
|---|---|
| | used for supportive analysis of the primary efficacy endpoint only. The PP population will not be analysed if this population comprises more than 95% or less than 50% of the ITT population. |
| | All the summary and analysis will be performed for both ITT population and Subset ITT population (2 to 6 years old). The ITT, Subset ITT and PP populations will be determined prior to unblinding of the study (except for the PD of incorrect treatment container ID, which can be determined only after unblinding). |
| Hypothesis | No formal hypothesis test will be done in this study. All the results from analysis modelling are for descriptive purpose. |
| Primary<br>Analyses | The mean change from baseline over the first 2 weeks treatment period in daily rTNSS (rhinorrhea, nasal congestion, nasal itching, and sneezing) will be analyzed using the method of pairwise comparison of treatment groups (active vs. placebo) with analysis of covariance (ANCOVA) adjusting for baseline daily rTNSS, classification of AR (IAR or PER), age (as continuous variable), gender, and treatment. |
| Secondary<br>Analyses | Regarding the secondary analyses for diary card endpoints (rTOSS over 2 weeks, rTOSS and rTNSS over 4 weeks), the analysis method will be the same as the primary efficacy analysis. |
| | Overall evaluation of response to therapy for subjects will be summarized, and analysed using logistic regression adjusting for age (as continuous variable), gender, classification of AR (IAR or PER), and treatment. |
| | ANCOVA model adjusting for baseline nasal finding score by anterior rhinoscopy, classification of AR (IAR or PER), age (as continuous variable), gender, and treatment will be used to analyse nasal finding score by anterior rhinoscopy. |
| | ANCOVA model adjusting for classification of AR (IAR or PER), age (as continuous variable), gender, and treatment will be used to analyse the mean rescue-free days over the first 2 weeks and over the 4 weeks treatment. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 15-JAN-2016).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To establish the efficacy of FFNS 55 µg and 110 µg QD versus vehicle placebo nasal spray in paediatric subjects (ages 2 to 12 years old) with | Mean change from baseline over the first 2 weeks treatment period in daily, reflective total nasal symptom scores (rTNSS) in subjects ages 2 to 12 years old Secondary Endpoints |
| AR | Overall evaluation of response to therapy (evaluated on a 7-point categorical scale) after the first 2 weeks treatment (day15) |
| | <ul> <li>Mean change from baseline of intranasal finding score by<br/>anterior rhinoscopy at the first 2 weeks (day 15)</li> </ul> |
| | <ul> <li>Mean change from baseline over the first 2 weeks<br/>treatment period in the daily, reflective total ocular<br/>symptoms score (rTOSS)</li> </ul> |
| | Rescue loratadine use (mean rescue-free days) over the first 2 weeks treatment period |
| | <ul> <li>Mean change from baseline over the 4 weeks treatment<br/>period in daily rTNSS</li> </ul> |
| | <ul> <li>Overall evaluation of response to therapy after 4 weeks<br/>treatment period (day 29)</li> </ul> |
| | The mean change from baseline of intranasal finding<br>score by anterior rhinoscopy at the end of treatment (day<br>29) |
| | Mean change from baseline over the 4 weeks treatment period in the daily rTOSS |
| | Rescue loratadine use (mean rescue-free days) over the entire 4 weeks treatment period |
| Secondary Objectives | Safety Endpoints |
| To investigate the safety of FFNS 55 µg and 110 µg QD versus vehicle placebo nasal spray in paediatric | <ul> <li>Frequency and type of clinical adverse events</li> <li>Results of clinical laboratory tests (haematology, chemistry and urinalysis)</li> </ul> |
| subjects (ages 2 to 12 years old) with AR | <ul> <li>Results of physical and nasal examination</li> <li>Vital signs (systolic and diastolic blood pressures, pulse rate and respiratory rate)</li> </ul> |

# 2.3. Study Design



# 2.4. Statistical Hypotheses

The study is designed to provide an estimated mean treatment difference between active drug groups and placebo group in primary efficacy endpoint, change from baseline of daily rTNSS over the first 2 weeks treatment period. No formal hypothesis test will be done. All the results from analysis modeling are for descriptive purpose.

The primary comparisons of interest between treatment groups are:

FFNS 55 µg vs Placebo

FFNS 110 µg vs Placebo

As a supportive comparison, the pooled active drug groups (low and high-dose) will be compared with placebo.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No interim analysis is planned.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled | Comprise of all subjects, for whom a record exists on the study database, including screen/run-in failures and any subject who was not screened but experienced an SAE between the date of informed consent and the planned date of the Screening Visit. | Reporting subject disposition,<br>reasons for screen/run-in<br>failures, and inclusion,<br>exclusion and randomization<br>criteria deviations and SAEs<br>for non-randomized subjects |
| Intent-To-Treat | Comprise of all randomized subjects<br>who received at least one dose of study<br>treatment. | The primary analysis population for efficacy analysis |
| | Subjects will be analyzed according to | Safety analysis |
| | the treatment they were randomly assigned to. | Summary of demographic and baseline |
| | Any subject who receives a treatment<br>randomization number will be<br>considered to have been randomized. | |
| | The decision to exclude a subject from<br>the ITT Population will be made prior to<br>breaking the blind. | |
| Subset Intent-<br>To-Treat (2 to 6 years old) | Comprise of all subjects in the ITT Population aged ≥2 to ≤6 years old | The analysis population for efficacy and safety on subjects aged ≥2 to ≤6 years |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | | old • Summary of demographic and baseline on subjects aged ≥2 to ≤6 years old |
| Per-Protocol | Comprise of all randomized subjects in<br>ITT population who do not have any full<br>protocol deviations. | The supportive analysis population for primary efficacy endpoint only. |
| | Subjects identified as partial protocol violators will be included in the PP Population but will have their data excluded from PP analyses from the time of violation onwards. | The PP population will not be analyzed if this population comprises more than 95% or less than 50% of the ITT population. |
| | The definition of full and partial violations will be included in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population). | |
| | The decision to exclude a subject from<br>the PP Population or a subject's data<br>from PP analyses will be made prior to<br>breaking the blind (except the PD of<br>incorrect treatment container ID, which<br>only can be defined after unblinding). | |

# 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.


201492

• A separate summary and listing of all inclusion/exclusion/randomisation criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion/randomisation page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Treatment States and Phases |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |
| 11.9 | Appendix 9: Multicentre Studies |
| 11.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 11.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 11.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| 11.13 | Appendix 13: Abbreviations & Trade Marks |
| 11.14 | Appendix 14: List of Data Displays |
| 11.15 | Appendix 15: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Intent-To-Treat population and subset Intent-To-Treat population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Summary of Screening Subject Disposition | Y | | |
| Reasons for Exclusion from the Per Protocol Population | Υ | | Υ |
| Number of Subjects by Centre | Υ | | |
| Subject Accountability: End of Study Record | Υ | | |
| Subject Withdrawals: End of Study Record | | | Υ |
| Number of Subjects at Each Visit | Υ | | |
| Protocol Deviations | | | |
| Inclusion/ Exclusion/Randomisation Criteria Deviations | Υ | | Υ |
| Important Protocol Deviations | Υ | | Υ |
| Date of and Reason for Breaking Treatment Blind During | | | Υ |
| the Study | | | Ī |
| Demography | | | |
| Demographics Characteristics | Υ | | Υ |
| Medical Condition | | | |
| Summary of Allergy History | Υ | | Υ |
| Summary of Baseline Nasal Symptom Scores | Υ | | |
| Summary of Medical Conditions | Υ | | Υ |
| Concomitant Medication | | | |
| Relationship between ATC Level 1, Ingredient and | Υ | | |
| Verbatim Text | Ī | | |
| Summary of Concomitant Medications | Υ | | Υ |
| Treatment Compliance | _ | | |
| Treatment compliance | Υ | | |

### NOTES:

- Y = Yes display generated.
- All summaries tables will be presented by treatment group.

### 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Efficacy Analyses

# 7.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the Intent-To-Treat population (of primary interest), PP population (supportive if appropriate) and the subset ITT-2 to 6 years old population (supportive), unless otherwise specified.

Table 3 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | | | - 1 | Absol | ute | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sta | ts Ana | lysis | Sun | mary | Indiv | ridual | Stats Analysis | | | Summary | | Individual | |
| | Τ | F | L | Т | F | F | L | Т | F | Г | Т | F | F | L |
| <b>Primary Efficacy Analys</b> | Primary Efficacy Analyses | | | | | | | | | | | | | |
| Baseline Daily | | | | Υ | | | Υ | | | | | | | |
| Reflective Total Nasal | | | | | | | | | | | | | | |
| Symptom Scores | | | | | | | | | | | | | | |
| Daily Reflective Total | | | | Υ | | | Υ | | | | Υ | Υ | | Υ |
| Nasal Symptom Scores | | | | | | | | | | | | | | |
| Mean Daily Reflective | | | | Υ | | | Υ | Υ | | | Υ | Υ | | Υ |
| Total Nasal Symptom | | | | | | | | | | | | | | |
| Scores over Each Week | | | | | | | | | | | | | | |
| Mean Daily rTNSS over | | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| the First 2 Weeks | | | | | | | | | | | | | | |
| Mean Daily rTNSS over | | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| the 4 Weeks Treatment | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.

### 7.1.2. Planned Efficacy Statistical Analyses

### **Primary Statistical Analyses**

### Endpoint(s)

- Mean change from baseline of Daily rTNSS over Each Week
- Mean change from baseline of Daily rTNSS over the First 2 Weeks
- Mean change from baseline of Daily rTNSS over the 4 Weeks

### **Model Specification**

- Endpoints will be statistically analyzed using analysis of covariance (ANCOVA) model adjusting for baseline daily rTNSS, classification of AR (IAR or PER), age (as continuous variable), gender and treatment.
- No imputations will be performed on missing daily diary data.

# **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

### **Model Results Presentation**

- LS mean change from baseline values for each treatment group will be presented with their associated standard errors.
- Estimated treatment differences along with corresponding 95 % confidence intervals (CIs) and p-values will be presented for the treatment comparisons.

### **Sensitivity and Supportive Statistical Analyses**

 The summaries, figures and analysis detailed in Section 7.1.1 (Overview of Planned Efficacy Analyses) and above primary statistical analyses, will be repeated for the PP population and subset ITT (2 to 6 years old) population.

### 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Efficacy Analyses

# 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the Intent-To-Treat population (of primary interest), and the subset ITT-2 to 6 years old population (supportive), unless otherwise specified.

Table 4 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| Endpoint | | Absolute | | | | | | | Cl | hange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sumr | nary | Indiv | idual | Stats Analysis | | | Sum | mary | Indiv | idual |
| | Τ | F | L | Τ | F | F | L | Τ | F | L | Т | F | F | L |
| Daily Reflective Total | | | | Υ | | | Υ | | | | Υ | | | Υ |
| Ocular Symptom | | | | | | | | | | | | | | |
| Scores | | | | | | | | | | | | | | |
| Mean Daily Reflective | | | | Υ | | | Υ | Υ | | | Υ | Υ | | Υ |
| Total Ocular Symptom | | | | | | | | | | | | | | |
| Scores over Each | | | | | | | | | | | | | | |
| Week | | | | | | | ., | ., | | | ., | | | |
| Mean Daily rTOSS | | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| over the First 2 Weeks | | | | \ | | | \/ | \/ | | | | | | |
| Mean Daily rTOSS | | | | Υ | | | Y | Υ | | | Υ | | | Υ |
| over the 4 Weeks | | | | | | | | | | | | | | |
| Treatment Overall Evaluation of | Υ | | | Υ | | | Υ | | | | | | | |
| Response to Therapy | ľ | | | ľ | | | Y | | | | | | | |
| after the First 2 Weeks | | | | | | | | | | | | | | |
| and 4 Weeks | | | | | | | | | | | | | | |
| Treatment | | | | | | | | | | | | | | |
| Intranasal Finding | | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| Score by Anterior | | | | ' | | | | | | | • | | | |
| Rhinoscopy at the First | | | | | | | | | | | | | | |
| 2 Weeks and 4 Weeks | | | | | | | | | | | | | | |
| Treatment | | | | | | | | | | | | | | |
| Rescue Loratadine | Υ | | | Υ | | | Υ | | | | | | | |
| Use (Mean Rescue- | | | | | | | | | | | | | | |
| free Days) over the | | | | | | | | | | | | | | |
| First 2 Weeks and 4 | | | | | | | | | | | | | | |
| Weeks Treatment | | | | | | | | | | | | | | |
| NOTES · | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

All the tables will be presented by treatment group.

# 8.1.2. Planned Efficacy Statistical Analyses

### **Primary Statistical Analyses**

### Endpoint(s)

- Overall evaluation of response to therapy (evaluated on a 7-point categorical scale) after the first 2 weeks treatment (day 15)
- The mean change from baseline of study intranasal finding score by anterior rhinoscopy at the first 2 weeks treatment (day 15)
- Mean change from baseline over the first 2 weeks treatment period in the daily reflective total ocular symptoms score (rTOSS)
- Rescue loratadine use (mean rescue-free days) over the first 2 weeks treatment period
- Overall evaluation of response to therapy after 4 weeks treatment period (day 29)
- The mean change from baseline of intranasal finding score by anterior rhinoscopy at the end of treatment (day 29)
- Mean change from baseline over the 4 weeks treatment period in the daily rTOSS
- Rescue loratatine use (mean rescue-free days) over the entire 4 weeks treatment period

### **Model Specification**

- Overall evaluation of response to therapy (evaluated on a 7-point categorical scale) after the first 2 weeks treatment and 4 weeks will be analyzed using a logistic regression.
- Terms fitted in the logistic regression model will be included: Treatment, classification of AR (IAR or PER), gender, age (as continuous variable).
- For the Rescue loratadine use (mean rescue-free days) will be analyzed using an ANCOVA analysis
- Terms fitted in the ANCOVA model will be included:

Fixed Categorical Covariates :Treatment, classification of AR (IAR or PER),

gender

Fixed Continuous Covariates : age

- For the secondary endpoints of rTOSS and nasal finding score by anterior rhinoscopy will be analyzed using an ANCOVA analysis.
- Terms fitted in the ANCOVA model will be included:

Fixed Categorical Covariates :Treatment, classification of AR (IAR or PER),

gender

Fixed Continuous Covariate : Baseline value of endpoint, age

### **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For the ANCOVA model
  - ✓ LS means values for each treatment group will be presented with their associated standard errors.
  - ✓ Estimated treatment differences along with corresponding 95% CIs and p-values will be presented for the treatment comparisons.
- For the logistic regression model
  - ✓ Frequencies and percentages for each treatment group will be presented with each category.
  - ✓ P-values will be presented for the treatment comparisons.

# 8.2. Safety Analyses

# 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the Intent-To-Treat and subset Intent-To-Treat (2 to 6 years old) population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint | | Abs | olute | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | Individual | | Summary | | Individual |
| | T | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | Y | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| On-Treatment AEs | Υ | | | | | | | |
| Post-Treatment AEs | Υ | | | | | | | |
| AEs with Incidence | Υ | | | | | | | |
| Rate >3% in Any | | | | | | | | |
| Treatment Group and | | | | | | | | |
| More Common than | | | | | | | | |
| Placebo During the | | | | | | | | |
| Treatment Period | | | | | | | | |
| On-treatment Drug- | Y | | | Υ | | | | |
| Related AEs | | | | | | | | |
| Relationship of Primary | Υ | | | | | | | |
| SOC, Preferred Term | | | | | | | | |
| and Verbatim | | | | | | | | |
| All AEs | | | | Υ | | | | |
| Serious Adverse Event | s | | | | | | | |
| SAEs | Υ | | | Υ | | | | |
| Adverse Events Leadin | g to Disc | ontinuatio | n of Study | Treatmen | t and Othe | er Signific | ant Adver | se |
| Events | | | | | | | | |
| AEs Leading to | Y | | | Υ | | | | |
| Discontinuation of | | | | | | | | |
| Study Treatment | | | | | | | | |
| Nasal examination | | | | | | | | |
| Nasal examination | Y | | | Υ | | | | |
| results by visit | | | | | | | | |
| Shift from baseline | Υ | | | | | | | |
| Abnormal nasal | | | | Υ | | | | |
| examination results | | | | | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Υ | | | Υ | Υ | | | |
| Clinical Chemistry | Υ | | | | | | | |
| values outside the | | 1 | ] | | | | | 1 |
| values outside the | | | | | | | | |

| Endpoint | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| ' | Sum | mary | Indiv | /idual | | mary | Individual | |
| | T | F | F | L | Т | F | F | L |
| Clinical Chemistry | Υ | | | | | | | |
| Shifts from Baseline to | | | | | | | | |
| Endpoint | | | | | | | | |
| Subjects with at Least | | | | Υ | | | | |
| One Abnormal Value | | | | | | | | |
| Post-Randomization in | | | | | | | | |
| Chemistry | | | | | | | | |
| Haematology | Υ | | | Υ | Y | | | |
| Haematology values | Υ | | | | | | | |
| outside the normal | | | | | | | | |
| range | | | | | | | | |
| Haematology Shifts | Υ | | | | | | | |
| from Baseline to | | | | | | | | |
| Endpoint Subjects with at Least | | | | Υ | | | | |
| One Abnormal Value | | | | I | | | | |
| Post-Randomization in | | | | | | | | |
| Haematology | | | | | | | | |
| Routine Urinalysis | Υ | | | Y | | | | |
| Vital Signs | ' | | | | | | | |
| Pulse Rate | Υ | | | | Υ | | | |
| Systolic Blood | Y | | | | Y | | | |
| Pressure | - | | | | | | | |
| Diastolic Blood | Υ | | | | Υ | | | |
| Pressure | | | | | | | | |
| Respiratory Rate | Υ | | | | Υ | | | |
| Temperature | Υ | | | | Υ | | | |
| 12-Lead ECG | | | • | | | | | • |
| QTc | Υ | | | | Υ | | | |
| PR Interval | Υ | | | | Υ | | | |
| Heart Rate | Υ | | | | Y | | | |
| ECG Findings | Υ | | | | | | | |
| ECG Abnormal | - | | | Y | | | | |
| Clinically Significant | | | | | | | | |

# NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.

# 9. OTHER STATISTICAL ANALYSES

No other statistical analysis is planned.

### 10. REFERENCES

Chinese Medical Association of Otorhinolaryngology, Head and Neck Surgery, Pediatric group. Chinese Guideline for Diagnosis and Treatment of AR in Pediatrics. Chin J Otorhinolaryngol Head Neck Surg. 2011;46:7-8.

GSK Document Number RM2004/00130/05 Investigator's Brochure for Intranasal Fluticasone Furoate. 15-DEC-2011.

ICH Expert Working Group, Statistical Principles for Clinical Trials, E9, 1998.

Ruchi, Gupta, Kevin B. Weiss,. The 2007 National Asthma Education and Prevention Program Asthma Guidelines: Accelerating Implementation and Facilitating Their Impact Children With Asthma. Pediatrics. 2009;123:S193-198.

Schoenwetter WF, Dupclay L, Appajosyula S, Botteman MF, Pashos CL. Economic impact and quality-of-life burden of allergic rhinitis. Curr Med Res Opin. 2004;20(3):305-317.

Wallace DV, Dykewicz MS, Bernstein DI, Blessing-Moore J, Cox L, Khan DA et al. The diagnosis and management of rhinitis: An updated practice parameter. J Allergy Clin Immunol. 2008;122:S1-84.

GlaxoSmithKline document number 2014N205225\_02. Study 201492: A Randomized, Doubled-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of Fluticasone Furoate Nasal Spray 55 µg and 110 µg for 4 Weeks in Chinese Pediatric Subjects Ages 2 to 12 years with Allergic Rhinitis. Effective Date: 15-Jan-2016

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Assessment Windows |
| Section 11.4 | Appendix 4: Treatment States & Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 11.9 | Appendix 9: Multicentre Studies |
| Section 11.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 11.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 11.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 11.14 | Appendix 14: List of Data Displays |
| Section 11.15 | Appendix 15: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

### 11.1.1. Exclusions from Per Protocol Population

Protocol deviations identified here are those considered to affect the primary outcome of the study. All decisions on whether to exclude a subject from analysis will be made prior to breaking the blind, with the exception of subjects receiving incorrect treatment container. If, after breaking the blind, the container was found to have contained the correct randomised treatment, no data will be excluded from analyses.

# 11.1.2. Exclusions of Data from Per Protocol Analyses

Subjects with full protocol deviations identified below will be excluded from the PP population. Subjects with partial protocol deviations will generally be included in the PP population but have data excluded from PP analyses from the time of the deviation onwards.

#### 11.1.2.1 Inclusion/exclusion/randomisation Criteria Deviations

Failure of criteria will be considered a full protocol deviation as detailed in Table 6:

Table 6 Inclusion/exclusion/randomisation criteria deviations considered to affect the primary outcome

| Reason for exclusion | Full protocol deviation considered to affect primary outcome |
|---|---|
| Inclusion criterion | |
| Informed consent | Yes |
| Outpatient | No |
| Gender | No |
| Age | No |
| Diagnosis of AR | Yes |
| Exposure | No |
| Ability to Comply with Procedures | Yes |
| Exclusion criterion | |
| Concomitant Medical Conditions | depends |
| Concomitant Medication | depends |
| Subjects Will Travel More Than 48<br>Hours During the Study may Cause<br>the Change of Allergen | No |
| Investigators or Sub-investigators<br>Consider that a Subject is Not<br>Eligible | Yes |
| Randomisation criterion | |
| On the morning of Visit 2, subjects must have nasal or/and ocular | Yes |

| Reason for exclusion | Full protocol deviation considered to affect primary outcome |
|---|---|
| symptoms | |
| Average of the last 8 rTNSS assessments (4 AM assessments, 4 PM assessments) over the consecutive four 24-hours periods prior to randomization must be ≥6 | Yes |
| Average of the 8 reflective nasal symptom assessments for congestion (4 AM assessments, 4 PM assessments) over the consecutive four 24-hour periods prior to randomization must be ≥2 | Yes |

# 11.1.2.2 Programmed or and Manual Checks to Identify Deviations

The data checks identified in Table 7 will be performed to further identify protocol deviations.

Table 7 Programmed or/and Manual checks

| Reason for exclusion | Check performed | Deviation Type |
|---|---|---|
| Compliance with treatment | Overall compliance < 80 % or > 120% | Full |
| Incorrect treatment | At any point | Partial; data excluded from start of incorrect treatment onwards |
| Blind broken | At any point | Partial; data excluded from date of breaking of blind |
| Meet the following withdrawal criteria defined in the protocol but not withdrawn - A subject is significantly non-compliant with the requirements of the protocol. | At any point | Partial; data excluded from date of PD happened. |
| Prohibited medication | At any point | Partial; data excluded from date of PD happened. |

removed since use of these drugs should not affect lung function.be excluded from PP analyses from the start of the disallowed medication onwards.be excluded from PP analyses from the start of the disallowed medication onwards

# 11.2. Appendix 2: Time & Events

# 11.2.1. Protocol Defined Time & Events<sup>1</sup>

| | | | Early | F . II . | | | |
|---|---|---|---|---|---|---|---|
| Procedure | 1 | 2 | withdraw | Follow up | | | |
| | | | Study Day | | | | |
| Visit window (of days) | -4 to -14 | 1 | 8±2 | 15±2 | 29±2 | | 5±2 days<br>after V5 or<br>EW |
| Informed consent <sup>2</sup> | Х | | | | | | |
| Subject number | Х | | | | | | |
| assignment | | | | | | | |
| Medical history | X | | | | | | |
| Verification of inclusion/exclusion criteria | Х | | | | | | |
| Skin testing / serum-<br>specific IgE test (if not<br>done within 12 months of<br>visit 1) | X | | | | | | |
| Clinical laboratory<br>tests[Randomisation] if<br>applicable | Х | | | | Х | Х | |
| 12-Lead electrocardiogram | Х | | | | Х | Х | |
| Verification of randomized criteria | | Х | | | | | |
| Randomization number assignment | | Х | | | | | |
| Dispense double-blind study drug | | Х | | | | | |
| Dispense rescue loratadine | | Х | X3 | X3 | | | |
| Nasal spray technique education | | Х | Х | X | | | |
| Collect study drug | | | | | Х | Х | |
| Review screening diary <sup>4</sup> | | Х | | | | | |
| Review medical problem/medication dairy <sup>5</sup> | | Х | Х | X | Х | Х | |
| Compliance assessment | | | Х | Х | Х | Х | |
| Review treatment diary <sup>4</sup> | | | Х | Х | Х | Х | |
| Anterior rhinoscopy | | Х | Х | Х | Χ | Х | |
| Investigator assess overall response to therapy | | | | Х | Х | Х | |
| Vital Signs | X | | | | Х | Х | |
| Nasal examination | X | Х | Х | X | X | X | |
| Physical examination | X | | | , | X | X | |
| • | | | | | <u> </u> | | ., |
| AE/SAE review | <b>X</b> 6 | ←==== | :======= | ======= | ===== | X | X |

| Procedure | | , | Early | | | | |
|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 | withdraw | Follow up |
| | | | Study Day | I. | | | |
| Visit window (of days) | -4 to -14 | 1 | 8±2 | 15±2 | 29±2 | | 5±2 days<br>after V5 or<br>EW |
| Concomitant medication review | | <b>←===</b> | ======== | Х | Х | | |

- 1. Parent/guardian will record the symptom diary instead of subjects for all ages. The involvement of the parent/guardian in assessing and rating rhinitis symptoms may vary per subject. While it may not always be possible, the preference is for a consistent level of parent/guardian involvement throughout the study.
- 2. Informed Consent must be obtained prior to performing any Visit 1 procedures.
- 3. The dispense will depends on as needed.
- 4. The diary collects rTNSS, rTOSS, rescue usage and study medication usage.
- 5. The diary collect any medical problem (other than AR) and any medications used.
- 6. Serious AEs will be recorded from the time the consent form is signed until the follow-up visit. All AEs will be recorded from the start of study treatment until the follow-up visit.

# 11.3. Appendix 3: Assessment Windows

Assessment windows for the scheduled study visits are as follows:

Visit 1 Screening (4 to 14 days prior to randomization)

Visit 2 Randomization (Day 1)

Visit 3 (8  $\pm$  2 days after Visit 2, Week 1)

Visit 4 (15  $\pm$  2 days after Visit 2, Week 2)

Visit 5 (29  $\pm$  2 days after Visit 2, Week 4)

Individual assessments collected outside of the assessment window of scheduled visits will be included in the analysis without adjustment. If multiple assessments were collected within the same assessment window, the last valid value prior to randomization was used as the baseline value and the first valid value was used for all post-randomization visits.

will still be included in all ITT analyses.

# 11.4. Appendix 4: Treatment States and Phases

### 11.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date ≥ Study Treatment Stop Date + 2 |

#### NOTES:

If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 11.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 11.4.2.1. Treatment States for Concomitant Medications Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Medication start date < Study Treatment Start Date |
| On-Treatment | Medication start date ≤ Study Treatment Stop Date and Medication stop date≥ Study Treatment Start Date |
| Post-Treatment | Medication stop date > Study Treatment Stop Date |

#### NOTES:

- A medication will be classed in every period of the study in which it was taken.
- For medications with partial start and stop dates or missing start/stop dates, the medication will be classed in every period of the study in which it could have been taken.
- If the study treatment stop date is missing then the medication will be considered to be On-Treatment.
- The answers to the questions "Taken Prior to Study?" and "Ongoing?" which are recorded on the eCRF will also be taken into consideration to determine if the medication was started pre-treatment or continued post-treatment. In each case, should the answers suggest a different classification than the dates, the medication will be summarised in all possible classifications (pre/on/post) in which it could conceivably have been taken.

#### 11.4.2.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop + 1 |
| Post-Treatment | AE Start Date > Study Treatment Stop Date + 1 |
| Onset Time | If Treatment Start Date > AE Onset Date |
| Since 1st Dose | = AE Onset Date - Treatment Start Date; |
| (Days) | If Treatment Start Date ≤ AE Onset Date |
| | = AE Onset Date - Treatment Start Date + 1 |
| | Missing otherwise. |

| Treatment State | Definition |
|---|---|
| Duration (Days) | AE Resolution Date - AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

### NOTES:

- If the AE onset date is missing or partial then the AE will be considered on-treatment unless there is evidence to the contrary (e.g. the month of the onset date is present and is less than the month of the first dose of study treatment).
- AEs reported by subjects who did not receive treatment will be considered pre-treatment.
- Any SAEs for screen failures, run-in failures or subjects who were randomised but did not receive treatment will be classified as pre-treatment SAEs.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

### 11.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | ng |
| Code | Description | Description | Order [1] |
| Α | GW685698 55 µg QD | FF 55 µg QD | 2 |
| В | GW685698 110 μg QD | FF 110 µg QD | 3 |
| D | Pooled GW685698 Groups | FF 55/110 µg QD | 4 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

#### 11.5.2. Baseline Definition & Derivations

#### 11.5.2.1. Baseline Definitions

For all endpoints (except diary card) the baseline value will be the latest pre-dose assessment.

The baseline period for diary card endpoints is defined as 4 days prior to randomization, including the AM symptom assessment on the randomization (i.e., treatment initiation) date.

#### 11.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline Value |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- If either the baseline or on-treatment value is missing then the change from baseline will be set to missing.
- The change from baseline will not be calculated for baseline records or records prior to baseline.

# 11.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The version 9.2 of SAS software will be used. | |
| Reporting Area | |
| HARP Server | Not applicable since this is a CRO study |
| HARP Area | Not applicable since this is a CRO study |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

| Reporting Process |
|---------------------------------------------------------------------------|
| QC Spreadsheet Not applicable since this is a CRO study |
| Analysis Datasets |
| Analysis datasets will be created according to GSK A&R dataset standards. |
| Generation of RTF Files |
| RTF and PDF files will be generated. |

### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|--------------------------------|--------------------------------------------|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N. n. frequency. % |

# CONFIDENTIAL

201492

# Reporting Standards

# **Graphical Displays**

• Refer to IDSL Statistical Principals 7.01 to 7.13.

# 11.6. Appendix 6: Derived and Transformed Data

### 11.6.1. General

# **Multiple Measurements at One Time Point**

- The last valid value prior to randomization will be used as the baseline value (except diary card)
- The first valid measurement will be used for post-randomization visits in any derivation of summary statistics but if listed, all data will be presented.

### **Study Day**

When calculating the number of days relative to the date of randomization (i.e., treatment start date), the date of randomization will be counted as Day 1. Study day will be calculated as follows:

- Date of the event = Missing 
  → Study Day = Missing
- Date of the event < Start of treatment date → Study Day = Date of the event Start of treatment date
- Date of the event ≥ Start of treatment date → Study Day = Date of the event (Start of treatment date) + 1

# Date of Completion/Withdrawal

The date of completion/withdrawal will be derived as follows:

- For subjects who complete the last on-treatment study visit, the date of completion/withdrawal will be the date of that visit (Visit 5).
- For subjects who withdraw from the study, the date of completion/withdrawal will be the latest of the date of the last attended scheduled clinic visit (excluding follow-up), the date of the EW visit (if present) and the last dose date.

### 11.6.2. Study Population

#### **Demographics**

# Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
  - Age will be calculated based on the screening date.
- Birth date will be presented in listings as 'DDMMMYYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### Treatment Compliance Based on Subject Diary Card

The number of doses of study drug taken during the double-blind treatment period will be estimated based on information recorded by the subject on the diary card. Subjects will document their study

### Treatment Compliance Based on Subject Diary Card

medication administration/compliance on the diary card by answering the question "Did you spray 2 sprays of your medication in each nostril?" Each occurrence of "yes" in response to this question will count as one dose of study medication. Percent treatment compliance will be calculated for each subject as follows:

% Treatment Compliance = # of doses used x 100%, where expected # of doses used

- # of doses used = sum of the "yes" responses to the question "Did you spray 2 sprays of your medication in each nostril?" for all days on treatment
- expected # of doses used = # of days on treatment.

Overall compliance will be categorised as follows:

< 80%  $\geq 80\%$  to  $\leq 120\%$ >120%.

### 11.6.3. Safety

### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = (Treatment Stop Date –Treatment Start Date) + 1
- If a subject's **treatment** stop date is missing it will be assumed to be date of the study discontinuation/completion. If the study discontinuation/completion date is also missing then the extent of exposure will be set to missing.
- If a subject's **treatment** start date is missing then it will be assumed to be their Day 1 visit date.

# **Laboratory Parameters**

- The baseline value for a parameter will be the most recent recorded value for that parameter before dosing on Day 1.
- Laboratory data values will be classified as 'low', 'normal' or 'high' with reference to normal ranges.
- Laboratory data (haematology, chemistry, and urinalysis) will be collected during Visit 1
  (Screening) and Visit 5 (Week 4) / Early Withdrawal. The laboratory data will be summarized by
  visit. The number and percentage of subjects with laboratory values outside the normal range
  will be summarized by study visit for each laboratory analyte.
- Shift tables will summarize post-treatment flag values [low (L), normal (N), or high (H)] for each analyte, relative to their baseline flag values. Laboratory values are flagged as "low" if they are less than the lower limit of the normal range, "normal" if they are within the normal range and "high" if they are above the upper limit of the normal range. Baseline is defined as the last laboratory values captured prior to randomization [i.e., at Visit 1 or, where applicable, a repeat assessment performed prior to administration of the first dose of study medication at Visit 2

#### **Laboratory Parameters**

(Randomization, Day 1)]. The endpoint is defined as the first post-treatment value (i.e. laboratory value collected at Visit 5 (Week 4) or withdrawal visit). Shift from baseline to endpoint (Week 4 / discontinuation) in laboratory value is categorized, for each laboratory analyte, as follows:

To High L to H, N to H

To Normal or No Change L to N, H to N, L to L, N to N, H to H

To Low N to L, H to L.

The number of subjects in each category will be summarized for each laboratory analyte.

 All laboratory values for subjects with at least one post-treatment laboratory value (Including repeat assessments) outside the normal range will be listed.

#### **Nasal Examinations**

- The baseline value for a nasal examination endpoint will be the most recent recorded value for that endpoint before dosing on Day 1.
- Nasal examinations will be collected during Visits 1-5 or Early Withdrawal. Summary statistics
  for mucosa, septum, secretions, nasal patency, size of any polyps and ulcers will be provided at
  Visit 1-5 or Early Withdrawal.
- A summary of change from baseline in nasal examinations at endpoint (Vsit5/Early Withdrawal) will be made.

### **Vital Signs**

- The baseline value for a vital sign endpoint will be the most recent recorded value for that endpoint before dosing on Day 1.
- Vital signs will be collected during Visit 1 (Screening) and Visit 5 (Week 4)/Early Withdrawal.
   Summary statistics for systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (beats/min), temperature (°C), and respiratory rate (breaths/min) will be provided at baseline and Visit 5 or Early Withdrawal.
- A summary of change from baseline in vital signs at endpoint (Vsit5/Early Withdrawal) will be made.

#### 12-Lead ECG

- The baseline value for an ECG endpoint will be the most recent recorded value for that endpoint before dosing on Day 1.
- Twelve-lead ECGs will be performed at Visit 1 (Screening) and Visit 5 (Week 4)/Early Withdrawal. ECG results of "normal", "abnormal, not clinically significant (NCS)", and "abnormal, clinically significant (CS)" will be summarized at baseline and Visit 5 or Early Withdrawal.
- A listing of subjects with abnormal clinically significant ECG evaluations and/or clinically significant change(s) in ECG evaluations will be provided.

### 11.6.4. Efficacy

# Calculation of Baseline, Treatment Period, and Weekly Means for Symptom Scores

- For all diary-based efficacy assessments, the date of randomization (i.e., treatment start date)
   will be used as the reference date in defining the baseline and treatment periods.
- The baseline period for diary card endpoints is defined as 4 days prior to randomization, including the AM symptom assessment on the randomization (i.e., treatment initiation) date. For AM assessments, the baseline period includes the date of randomization and the 3 consecutive days prior to randomization. For PM assessments, the baseline period includes the 4 consecutive days prior to randomization. Baseline values for symptom scores are defined as the mean of the non-missing values for each symptom score during the baseline period.
- The first 2-week treatment period is defined as the first 14 dosing (24-hour) days after randomization. For the AM symptom assessments, the treatment period includes the first 14 consecutive days after the date of randomization. For the PM assessments, the treatment period includes the date of randomization and the 13 consecutive days following randomization. Treatment period values for symptom scores are defined as the mean of the non-missing values for each symptom score during the treatment period. No imputations will be performed on missing daily diary data.
- The mean change from baseline over the first 2 weeks/4 weeks of the treatment period in symptom scores (daily, AM, or PM) will be calculated as the subject's first 2- week/4-week treatment period mean minus the baseline period mean.
- Weekly values for symptom scores are defined in the same manner as the treatment period values (i.e., the mean of the non-missing values for each symptom score during a given 7-day week).

### Calculation of Total Nasal Symptom Scores (TNSS)

• The TNSS for each assessment time point is defined as the sum of the 4 individual nasal symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, and will range from 0 to 12. Each of the 4 individual nasal symptoms is evaluated by the subject using a 4-point (0 to 3) categorical scale and recorded on a diary card. The reflective scores (i.e., rTNSS) are ratings of the severity of symptoms over the previous 12 hours and are performed in the AM and PM. Daily (i.e., during one dosing interval) reflective scores are defined as the average of the PM reflective scores and the AM reflective scores of the next day prior to the AM dosing. For example, the Day 1 rTNSS will be computed as [(PM rTNSS) Day1, first day of dosing + (AM rTNSS) Day2, prior to second dosing]/2. And the Day 28 rTNSS will be computed as [(PM rTNSS) Day 29, last clinic visit]/2.
# 11.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

### 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as on completion of final on-treatment clinic visit (Visit 5).</li> <li>Withdrawn subjects will not be replaced in the study.</li> </ul> |
| | <ul> <li>All available data from subjects who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures,<br/>unless otherwise specified.</li> </ul> |
| | • In general, the minimum data required will be a baseline evaluation (if baseline is required for the analysis) and at least one post-baseline evaluation. |
| | <ul> <li>If a subject withdraws at a scheduled treatment visit, then any data collected at<br/>that visit associated with scheduled visit procedures will be used (under the<br/>scheduled visit assignment) in all summaries and analyses wherever possible.</li> </ul> |
| | Early withdrawal data will be included in relevant listing. |

## 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | • For efficacy endpoints, missing data is expected to arise mainly from subjects missing complete visits or time points. If for a given subject at a given assessment time (i.e., AM or PM) any of the 4 individual symptom scores are missing, then the TNSS will be considered missing for that assessment time. If one, but not both, of the AM and PM TNSS is missing for a given day (i.e., a dosing interval during the treatment period), the non-missing TNSS for that day will used as the daily TNSS for that day. |
| | <ul> <li>The amount of occasional missing data for covariates included in the statistical<br/>analysis is expected to be minimal. Missing data will not be imputed.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.7.2.1. Handing of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

## 11.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | Tartan actor or arry comocimicant moderations recorded in the erri vin se |
| Adverse<br>Events | , , |

## 11.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|------------------------------|-----------------------------------|
| ANCOVA | Missing data will not be imputed. |
| Logistic regression Analysis | Missing data will not be imputed. |

# 11.8. Appendix 8: Values of Potential Clinical Importance

Not applicable

# 11.9. Appendix 9: Multicentre Studies

This study was planned to be conducted in China. Approximately 12 investigative centres are expected to participate in the study. It is expected that most of investigational centres will have a small number of subjects, 10 subject per arm per centre. Given the small number of patients in each centre, centre will not be included as a covariate in the analysis models.

# 11.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

The details of covariates that will be used in statistical analyses have been clarified in Section 7 (Primary Statistical Analyses), 8 (Secondary Statistical Analyses).

For the modeling analysis on ITT-2 to ≤6 years old population, if the statistical model does not converge for all the covariates, sex, age will be dropped from the model. If the model still does not converge, then classification of AR (IAR or PER) will be further dropped. If the model still does not converge, the nonparametric ANCOVA method will be used. First ranking the observations from lowest to highest across all treatment groups, then using the ANCOVA methods on these ranks to test for significant treatment effect.

## 11.11. Appendix 11: Multiple Comparisons & Multiplicity

No multiplicity adjustments are necessary since no formal hypothesis test will be done.

# 11.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

#### 11.12.1. Statistical Analysis Assumptions

| Endpoint(s) | Mean change from baseline of daily rTNSS over each week |
|---|---|
| | <ul> <li>Mean change from baseline of daily rTNSS over the first 2 weeks treatment</li> </ul> |
| | <ul> <li>Mean change from baseline of daily rTNSS over the 4 weeks treatment</li> </ul> |
| Analysis | <ul> <li>ANCOVA</li> </ul> |

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored.
- The following SAS code will be used:

```
proc mixed data= adeff;
```

by week;

```
class treatment gender iarper;
```

model endpoint=treatment baseline gender age iarper;

lsmeans treatment / cl diff e om;

ods output lsmeans=lsmeans;

ods output diffs=diffs;

run;

| Endpoint(s) | • | Overall Evaluation of Response to Therapy |
|-------------|---|-------------------------------------------|
| Analysis | • | Logistic Regression Model |

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The following SAS code will be used:

```
proc logistic data=adeff descending;
```

by week;

class treatment (ref='1') gender iarper / param=ref;

```
model respond=treatment gender age iarper / clodds=wald expb;

ods output oddsratios=odds1

(where=(index(effect, 'TREATMENT')>0)

or index(effect, 'treatment')>0));

ods output parameterestimates=pval1

(keep=probchisq variable classval0

where=(variable in ('TREATMENT', 'treatment')));

ods output Type3=pval2

(where=(variable in ('TREATMENT', 'treatment')));

run;
```

# 11.13. Appendix 13: Abbreviations & Trade Marks

## 11.13.1. Abbreviations

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| AR | Allergic Rhinitis |
| BUN | Blood Urea Nitrogen |
| CPK | Creatinine Phosphokinase |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| FF | Fluticasone Furoate |
| IA | Interim Analysis |
| IAR | Intermittent Allergic Rhinitis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| INR | International Normalized Ratio |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| PER | Persistent Allergic Rhinitis |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QD | Quaque Die |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RBC | Red Blood Cells |
| SAC | Statistical Analysis Complete |
| SD | Standard deviation |

| Abbreviation | Description |
|--------------|------------------------------|
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TOSS | Total Ocular Symptom Score |
| TNSS | Total Nasal Symptom Score |
| WBC | White Blood Cells |

## 11.13.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RAMOS |
| Randall |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

## 11.14. Appendix 14: List of Data Displays

### 11.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.31 | |
| Efficacy | 2.1 to 2.22 | 2.1 to 2.10 |
| Safety | 3.1 to 3.53 | |
| Section | Listings | |
| ICH Listings | 1 to 15 | |
| Other Listings | 16 to 2 | 21 |

#### 11.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|------------|---------|
| Study Population | | 1.12 | |
| Efficacy | | | 20, 21 |
| Safety | | 3.26, 3.27 | |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 11.14.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 11.14.4. Study Population Tables

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 1.01. | All Subjects<br>Enrolled | ffr30008-01-body-csr<br>Table 6.1 | Summary of Screening Subject Disposition | | SAC [1] |
| 1.02. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.3 | Number of Subjects by Centre | | SAC [1] |
| 1.03. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.5 | Summary of Subject Accountability: End of Study Record | | SAC [1] |
| 1.04. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.5 | Summary of Subject Accountability: End of Study Record | | SAC [1] |
| 1.05. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.12 | Summary of Number of Subjects at Each Visit | | SAC [1] |
| 1.06. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.12 | Summary of Number of Subjects at Each Visit | | SAC [1] |
| 1.07. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.18 | Summary of Inclusion/Exclusion/Randomization Criteria Deviations | | SAC [1] |
| 1.08. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.18 | Summary of Inclusion/Exclusion/Randomization Criteria Deviations | | SAC [1] |
| 1.09. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.25 | Summary of Important Protocol Deviations | | SAC [1] |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 1.10. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.25 | Summary of Important Protocol Deviations | | SAC [1] |
| 1.11. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.25 | Summary of subjects excluded from the per-protocol population and reasons | | SAC [1] |
| 1.12. | All Subjects<br>Enrolled | Non-Standard: See appendix 15 | Summary of Analysis Populations | | SAC [1] |
| 1.13. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.37 | Summary of Demographic Characteristics | | SAC [1] |
| 1.14. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.37 | Summary of Demographic Characteristics | | SAC [1] |
| 1.15. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.49 | Summary of Allergy History | | SAC |
| 1.16. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.49 | Summary of Allergy History | | SAC |
| 1.17. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.56 | Summary of Baseline Nasal Symptom Scores | | SAC |
| 1.18. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.56 | Summary of Baseline Nasal Symptom Scores | | SAC |
| 1.19. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.60 | Summary of Past Medical Conditions | | SAC |
| 1.20. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.60 | Summary of Current Medical Conditions | | SAC |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable [Priority] |
| 1.21. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.60 | Summary of Past Medical Conditions | | SAC |
| 1.22. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.60 | Summary of Current Medical Conditions | | SAC |
| 1.23. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.62 | Relationship between ATC Level 1, Ingredient and Verbatim Text | | SAC |
| 1.24. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.63 | Summary of Concomitant Medications During the Pretreatment Period | | SAC |
| 1.25. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.63 | Summary of Concomitant Medications During the Pretreatment Period | | SAC |
| 1.26. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.64 | Summary of Concomitant Medications During the<br>Treatment Period | | SAC |
| 1.27. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.64 | Summary of Concomitant Medications During the<br>Treatment Period | | SAC |
| 1.28. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.64 | Summary of Concomitant Medications During the Post-treatment Period | | SAC |
| 1.29. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.64 | Summary of Concomitant Medications During the Post-treatment Period | | SAC |
| 1.30. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.80 | Summary of Treatment Compliance on Nasal Spray<br>Study Medication Based on Subject Diary Record | | SAC |
| 1.31. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 6.80 | Summary of Treatment Compliance on Nasal Spray<br>Study Medication Based on Subject Diary Record | | SAC |

#### CONFIDENTIAL

201492

# 11.14.5. Study Population Figures

No study population figure will be displayed.

# 11.14.6. Efficacy Tables

| Effica | cy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.01. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Daily Reflective Total Nasal Symptom Scores | Change Std Err to SD | SAC [1] |
| 2.02. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Daily Reflective Total Nasal Symptom Scores | Change Std Err to SD | SAC [1] |
| 2.03. | Per Protocol | ffr30008-01-body-csr<br>Table 7.1 | Summary of Daily Reflective Total Nasal Symptom Scores | Change Std Err to SD | SAC [1] |
| 2.04. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Daily Reflective Total Nasal Symptom Scores | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.05. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Daily Reflective Total Nasal Symptom Scores | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.06. | Per Protocol | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Daily Reflective Total<br>Nasal Symptom Scores | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.07. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Total Ocular Symptom Scores | Change Std Err to SD | SAC [1] |
| 2.08. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Total Ocular Symptom Scores | Change Std Err to SD | SAC [1] |
| 2.09. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Daily Reflective Total<br>Ocular Symptom Scores | Add a pooled active drug group (low and high-dose) column | SAC [1] |

| Effica | ıcy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Daily Reflective Total Ocular Symptom | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.11. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.11 | Analysis of Overall Evaluation of Response to Therapy after the first 2 weeks and 4 weeks treatment | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.12. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.11 | Analysis of Overall Evaluation of Response to Therapy after the first 2 weeks and 4 weeks treatment | Add a pooled active drug group (low and high-dose) column | SAC [1] |
| 2.13. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Intranasal Finding Score by Anterior Rhinoscopy | Change Std Err to SD | SAC |
| 2.14. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.1 | Summary of Intranasal Finding Score by Anterior Rhinoscopy | Change Std Err to SD | SAC |
| 2.15. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline of Intranasal Finding Score by Anterior Rhinoscopy | Add a pooled active drug group (low and high-dose) column | SAC |
| 2.16. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline of Intranasal Finding Score by Anterior Rhinoscopy | Add a pooled active drug group (low and high-dose) column | SAC |
| 2.17. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Rescue Loratadine Use (Mean Rescue-free Days) Over the First 2 Weeks and 4 Weeks Treatment | Add a pooled active drug group (low and high-dose) column | SAC |
| 2.18. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.2 | Analysis of Mean Change from Baseline in Rescue Loratadine Use (Mean Rescue-free Days) Over the First 2 Weeks and 4 Weeks Treatment | Add a pooled active drug group (low and high-dose) column | SAC |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.55 | Summary of Daily Reflective Total Nasal Symptom Scores Days 1-28 of the Treatment Period | | SAC |
| 2.20. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.55 | Summary of Daily Reflective Total Nasal Symptom Scores Days 1-28 of the Treatment Period | | SAC |
| 2.21. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 7.56 | Analysis of Mean Change from Baseline in Daily Reflective Total Nasal Symptom Scores Days 1-28 of the Treatment Period | | SAC |
| 2.22. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 7.56 | Analysis of Mean Change from Baseline in Daily Reflective Total Nasal Symptom Scores Days 1-28 of the Treatment Period | | SAC |

# 11.14.7. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.01. | Intent-to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Nasal Symptom Score Over the first 2 weeks Treatment Period | | SAC |
| 2.02. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Nasal Symptom<br>Score Over the first 2 weeks Treatment Period | | SAC |
| 2.03. | Per Protocol | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Nasal Symptom Score Over the first 2 weeks Treatment Period | | SAC |
| 2.04. | Intent-to-Treat | Intent-to-Treat ffr30008-01-body-csr Figure 7.2 Mean Change from Baseline in Daily Reflective Total Nasal Symptom Score Over the Entire Treatment Period | | SAC | |
| 2.05. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Nasal Symptom Score Over the Entire Treatment Period | | SAC |
| 2.06. | Per Protocol | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Nasal Symptom Score Over the Entire Treatment Period | | SAC |
| 2.07. | Intent-to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Ocular Symptom Score Over the first 2 weeks Treatment Period | | SAC |
| 2.08. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Ocular Symptom Score Over the first 2 weeks Treatment Period | | SAC |
| 2.09. | Intent-to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Ocular Symptom Score Over the Entire Treatment Period | | SAC |
| 2.10. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Figure 7.2 | Mean Change from Baseline in Daily Reflective Total Ocular Symptom Score Over the Entire Treatment Period | | SAC |

# 11.14.8. Safety Tables

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.01. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.1 | Summary of Extent of Exposure to Study Medication | | SAC |
| 3.02. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.1 | Summary of Extent of Exposure to Study Medication | | SAC |
| 3.03. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.5 | Relationship of Adverse Event System Organ Class, Preferred Term, and Verbatim Text | | SAC |
| 3.04. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.5 | Relationship of Adverse Event System Organ Class, Preferred Term, and Verbatim Text | | SAC |
| 3.05. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.7 | Summary of All Adverse Events During the Treatment Period | | SAC |
| 3.06. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.7 | Summary of All Adverse Events During the Treatment Period | | SAC |
| 3.07. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.10 | Summary of All Adverse Events During the Post-<br>Treatment Period | | SAC |
| 3.08. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.10 | Summary of All Adverse Events During the Post-<br>Treatment Period | | SAC |
| 3.09. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.8 | AEs with Incidence Rate >3% in Any Treatment Group and More Common than Placebo During the Treatment Period | | SAC |
| 3.10. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.8 | AEs with Incidence Rate >3% in Any Treatment Group and More Common than Placebo During the Treatment Period | | SAC |

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.11. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.16 | Summary of Drug-Related Adverse Events During the Study Period | | SAC |
| 3.12. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.16 | Summary of Drug-Related Adverse Events During the Study Period | | SAC |
| 3.13. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.19 | Summary of Serious Adverse Events During the Study Period | | SAC |
| 3.14. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.19 | Summary of Serious Adverse Events During the Study Period | | SAC |
| 3.15. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.21 | Summary of AEs Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | SAC |
| 3.16. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.21 | Summary of AEs Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | SAC |
| 3.17. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.32 | Definitions of Normal Ranges for Haematology Values | | SAC |
| 3.18. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.32 | Definitions of Normal Ranges for Chemistry Values | | SAC |
| 3.19. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.32 | Definitions of Normal Ranges for Urinalysis Values | | SAC |
| 3.20. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Haematology Data | | SAC |

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.21. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Haematology Data | | SAC |
| 3.22. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Chemistry Data | | SAC |
| 3.23. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Chemistry Data | | SAC |
| 3.24. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Urinalysis Data for Continuous Values | | SAC |
| 3.25. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.33 | Summary of Urinalysis Data for Continuous Values | | SAC |
| 3.26. | Intent-to-Treat | Non-Standard: See appendix 15 | Summary of Urinalysis Data for Categorical Values | | SAC |
| 3.27. | Subset Intent-<br>to-Treat | Non-Standard: See appendix 15 | Summary of Urinalysis Data for Categorical Values | | SAC |
| 3.28. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Haematology Data Outside the Normal Range | | SAC |
| 3.29. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Haematology Data Outside the Normal Range | | SAC |
| 3.30. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Chemistry Data Outside the Normal Range | | SAC |

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.31. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Chemistry Data Outside the Normal Range | | SAC |
| 3.32. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Urinalysis Data Outside the Normal Range | | SAC |
| 3.33. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.34 | Summary of Urinalysis Data Outside the Normal Range | | SAC |
| 3.34. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Haematology Shifts from Baseline to Endpoint | | SAC |
| 3.35. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Haematology Shifts from Baseline to Endpoint | | SAC |
| 3.36. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Chemistry Shifts from Baseline to Endpoint | | SAC |
| 3.37. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Chemistry Shifts from Baseline to Endpoint | | SAC |
| 3.38. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Urinalysis Shifts from Baseline to Endpoint | | SAC |
| 3.39. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.35 | Summary of Urinalysis Shifts from Baseline to Endpoint | | SAC |
| 3.40. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.42 | Summary of Nasal Examinations | | SAC |

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.41. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.42 | Summary of Nasal Examinations | | SAC |
| 3.42. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.43 | Summary of Nasal Examination Shifts from Baseline to Endpoint | | SAC |
| 3.43. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.49 | Summary of Nasal Examination Shifts from Baseline to Endpoint | | SAC |
| 3.44. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.70 | Summary of Vital Signs | | SAC |
| 3.45. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.70 | Summary of Vital Signs | | SAC |
| 3.46. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.71 | Summary of Change from Baseline in Vital Signs at Endpoint | | SAC |
| 3.47. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.71 | Summary of Change from Baseline in Vital Signs at Endpoint | | SAC |
| 3.48. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.70 | Summary of ECG | | SAC |
| 3.49. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.70 | Summary of ECG | | SAC |
| 3.50. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.71 | Summary of Change from Baseline in ECG at Endpoint | | SAC |

| Safet | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.51. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.71 | Summary of Change from Baseline in ECG at Endpoint | | SAC |
| 3.52. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.72 | Summary of ECG Findings | | SAC |
| 3.53. | Subset Intent-<br>to-Treat | ffr30008-01-body-csr<br>Table 8.72 | Summary of ECG Findings | | SAC |


201492

# 11.14.9. Safety Figures

No safety figure will be displayed.

# 11.14.10. ICH Listings

| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Study F | opulation | | | | |
| 1. | Per Protocol | ffr30008-01-body-csr<br>Table 6.2 | Listing of Reasons for exclusion from Per-Protocol | | SAC |
| 2. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.11 | Listing of Subject Withdrawals: End of Study Record | | SAC |
| 3. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.24 | Listing of Inclusion/Exclusion/Randomization Criteria Deviations | | SAC |
| 4. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 6.31 | Listing of Important Protocol Deviations | | SAC |
| Safety | | | | | |
| 5. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.4 | Listing of Exposure | | SAC |
| 6. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.14 | Listing of All Adverse Events | | SAC |
| 7. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.17 | Listing of Drug-Related Adverse Events During the Study Period | | SAC |
| 8. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.20 | Listing of Serious Adverse Events | | SAC |
| 9. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.22 | Listing of Adverse Events Leading to Discontinuation of Study Treatment | | SAC |
| 10. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.14 | Listing of All Adverse Events for On-treatment Adverse Events of Special Interest | | SAC |
| 11. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.36 | Listing of Laboratory Data for Subjects with at Least One Abnormal Value Post-Randomization in Haematology | | SAC |
| 12. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.37 | Listing of Laboratory Data for Subjects with at Least One Abnormal Value Post-Randomization in Chemistry | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 13. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.37 | Listing of Laboratory Data for Subjects with at Least One Abnormal Value Post-Randomization in Urinalysis | | SAC |
| 14. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.46 | Listing of Subjects with at Least One Abnormal Nasal Examination Result Post-Baseline | | SAC |
| 15. | Intent-to-Treat | ffr30008-01-body-csr<br>Table 8.73 | Listing of Subjects with at Least One Abnormal Clinically Significant and/or Clinically Significant Change in ECG from Baseline Classification | | SAC |

# 11.14.11. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable [Priority] |
| Study F | Population | | | | |
| 16. | Intent-to-Treat | ffr30008-01-body-<br>csr Table 6.34 | Listing of Subjects for Whom the Treatment Blind was Broken During the Study | | SAC |
| 17. | Intent-to-Treat | ffr30008-01-body-<br>csr Table 6.47 | Listing of Subject Demographic Characteristics | | SAC |
| 18. | Intent-to-Treat | ffr30008-01-body-<br>csr Table 6.55 | Listing of Allergy History | | SAC |
| 19. | Intent-to-Treat | ffr30008-01-body-<br>csr Table 6.73 | Listing of Concomitant Medications During the Study Period | | SAC |
| Efficac | y | | | | |
| 20. | Intent-to-Treat | Non-Standard: See appendix 15 | Listing of Daily Diary Endpoint | | SAC |
| 21. | Intent-to-Treat | Non-Standard: See appendix 15 | Listing of Derived Diary Endpoint | | SAC |

## 11.15. Appendix 15: Example Mock Shells for Data Displays

Protocol: 201492 (Fluticasone Furoate Nasal Spray) Page 1 of n

Population: All Subjects Enrolled

Table 1.12 Summary of Analysis Populations

| Analysis Populations | Placebo | FF 55 μg QD | FF 110 µg QD | Total |
|---|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Intent-to-Treat | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Subset Intent-To-Treat (2 to 6 years old) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Per-Protocol | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |

Protocol: 201492 (Fluticasone Furoate Nasal Spray)


Population: Intent-to Treat

Table 3.26 Summary of Urinalysis Data for Categorical Value

| Lab Test | Visit | | Placebo | FF 55 ug QD | FF 110 ug QD |
|---|---|---|---|---|---|
| | | | N=XXX | N=XXX | N=XXX |
| Urine Ketones (dipstick) | Screening | | XXX | XXX | XXX |
| | | Negative | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |
| | | + | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |
| | | ++ | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |
| | Endpoint | | XXX | XXX | XXX |
| | | Negative | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |
| | | + | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |
| | | ++ | XXX (XXX.X%) | XXX (XXX.X%) | XXX (XXX.X%) |

201492

Protocol: 201492 (Fluticasone Furoate Nasal Spray)


Population: Intent-to Treat

Listing 20 Listing of Daily Diary Endpoint

Treatment:Placebo

| Inv./Subj. | Study day | TNSS | TOSS | Rescue Medication |
|------------|-----------|------|------|-------------------|
| PPD | Baseline | XX | XX | |
| | Dayl | XX | XX | Y |
| | Day 28 | XX | XX | N |

Protocol: 201492 (Fluticasone Furoate Nasal Spray)


Population: Intent-to Treat

Listing 21 Listing of Derived Diary Endpoint

Treatment:Placebo

| Inv./Subj. | Study day | TNSS | TOSS | Rescue-free Day |
|------------|--------------|------|------|-----------------|
| PPD | Baseline | XX | XX | |
| | Week 1 | XX | XX | XX |
| | Week 4 | XX | XX | XX |
| | Over 2 Weeks | XX | XX | XX |
| | Over 4 Weeks | XX | XX | XX |